CLINICAL TRIAL: NCT05809284
Title: Determining the Mechanisms of Loss of CAR T Cell Persistence
Acronym: CARPERS
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: UCL/156503
Record Dates: First submitted 2023-03-03; First posted 2023-04-12 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Acute Lymphoblastic Leukemia With Failed Remission; Acute Lymphoblastic Leukemia Not Having Achieved Remission; Acute Lymphoblastic Leukemia, Pediatric; Acute Lymphoblastic Leukemia, Adult; Acute Lymphoblastic Leukemia, in Relapse
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Excess CAR-T samples following infusion Blood samples will be collected at protocol timepoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study of pediatric and young adult acute lymphoblastic leukaemia (ALL) patients treated with CD19 chimeric antigen receptor T-cells (CAR-T cells). The study will examine changes in CAR-T persistence over time and causal factors.

ELIGIBILITY:
Inclusion Criteria:

1. Children and young adults (age 25 years or younger) with relapsed/refractory ALL who are planned to receive licensed CD19-targeted CAR-T cell treatment (Tisagenlecleucel)
2. Written informed consent

Exclusion Criteria:

1. Patients receiving an alternate CD19-directed CAR T-cell product on a clinical trial
2. Any reason that in the opinion of the investigator, patients won't be able to adhere to the protocol

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is paediatric and young adult patients aged 25 or younger who have relapsed/refractory B-cell acute lymphoblastic leukaemia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to circulating CAR-T cell loss | Through study completion, until the last patient reaches 1 year post-infusion
  CAR-T persistence will be measured in the central lab from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Persis Amrolia, BSc,MBBS,PhD, Study Chair — UCL Institute of Child Health
Locations (3):
- United Kingdom (3):
  - Great Ormond Street Hospital, London
  - University College London Hospital, London
  - Royal Manchester Children's Hospital, Manchester